CLINICAL TRIAL: NCT04924322
Title: Age-dependent Heterogeneity in the Efficacy of Prophylaxis With Enoxaparin Against Catheter-associated Thrombosis in Critically Ill Children
Brief Title: Catheter-Related Early Thromboprophylaxis With Enoxaparin Studies
Acronym: CRETE
Status: Recruiting | Phase: Phase 2 / Phase 3 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: Children's Hospital Colorado (Other); Children's Hospital of Philadelphia (Other); BJC HealthCare (Other); Medical College of Wisconsin (Other); Children's of Alabama (Other); Golisano Children's Hospital (Unknown); Maria Fareri Children's Hospital (Unknown); Nationwide Children's Hospital (Other); New York Presbyterian Hospital (Other); Penn State University (Other); University of Iowa (Other); Johns Hopkins All Children's Hospital (Other); University of Oklahoma (Other); Eunice Kennedy Shriver National Institute of Child Health and Human Development (NICHD) (NIH); Children's Hospital of Illinois OSF Saint Francis Medical Center (Unknown); Hassenfeld Children's Hospital (Unknown)
Responsible Party: Principal Investigator, E. Vincent S. Faustino, Professor of Pediatrics (Critical Care), Yale University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: 2000030683; 1R01HD106326-01 (NIH)
Record Dates: First submitted 2021-06-07; First posted 2021-06-11 (Actual); Last update posted 2025-06-11 (Actual); Status verified 2025-06

CONDITIONS: Deep Venous Thrombosis
Keywords: child; critical illness; venous thromboembolism; enoxaparin; thrombin generation; bleed
MeSH Terms: conditions — Venous Thrombosis; Critical Illness; Venous Thromboembolism; Hemorrhage | interventions — Enoxaparin

STUDY DESIGN:
Intervention Model Description: Older children 1-17 years old and infants <1 year old will be randomized separately. Older children will be randomized 2:1 to prophylactic dose of enoxaparin or control stratified by age. Infants will be randomized 1:1:1 to therapeutic dose of enoxaparin with high or low anti-Xa target or control stratified by age.
Who Masked: Outcomes Assessor
Masking Description: The CRETE Studies are open-label with blinded endpoint. Systematic ultrasonographic assessment will be performed with the images blindly and centrally adjudicated.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Enoxaparin (Older Children Prophylactic) (Experimental): Prophylactic dose of enoxaparin for older children 1-17 years old.
  Interventions: Drug: Enoxaparin
- Control (Older Children) (No Intervention): Usual care without placebo for older children 1-17 years old.
- Enoxaparin (Infants Therapeutic High Anti-Xa Target) (Experimental): Therapeutic dose of enoxaparin for infants <1 year old with anti-Xa target of >0.5-1 IU/mL.
  Interventions: Drug: Enoxaparin
- Enoxaparin (Infants Therapeutic Low Anti-Xa Target) (Experimental): Therapeutic dose of enoxaparin for infants <1 year old with anti-Xa target of 0.2-0.5 IU/mL.
  Interventions: Drug: Enoxaparin
- Control (Infants) (No Intervention): Usual care without placebo for infants <1 year old.

INTERVENTIONS:
Drug: Enoxaparin — Enoxaparin is a LMWH produced from UFH that exerts its anticoagulant effects by binding to and inducing a conformational change in antithrombin to accelerate the inactivation of factor Xa and thrombin. Age-specified dose of enoxaparin will be administered within 24 hours after insertion of the CVC with the dose subsequently adjusted to pre-specified anti-Xa target.
  Other Names: Lovenox; Clexane
  Arms: Enoxaparin (Infants Therapeutic High Anti-Xa Target); Enoxaparin (Infants Therapeutic Low Anti-Xa Target); Enoxaparin (Older Children Prophylactic)

SUMMARY:
The goal of the CRETE Studies is to investigate the newly identified age-dependent heterogeneity in the efficacy of enoxaparin in reducing the risk of central venous catheter-associated deep venous thrombosis in critically ill children.

DETAILED DESCRIPTION:
Pediatric venous thromboembolism (VTE), which is predominantly deep venous thrombosis (DVT), is a top contributor to harm in hospitalized children. Its incidence increased by >300% in the past 2 decades. Critical illness and central venous catheter (CVC) are the most important risk factors for VTE in children. Among critically ill children, the risk of CVC-associated DVT (CADVT) is as high as 54% with 72% of cases in infants <1-year old. Pharmacologic prophylaxis is the most effective strategy against VTE in adults. However, due to paucity of age-appropriate evidence on its efficacy against CADVT, pharmacologic prophylaxis is uncommon in children. Extrapolation of evidence from adults is not appropriate because the hemostatic system changes significantly with age. The investigators recently completed a Bayesian phase 2b randomized clinical trial. In this trial, the investigators randomized critically ill children to early administration of prophylactic dose of enoxaparin, the most commonly used anticoagulant for prophylaxis, or usual care. Prophylaxis with enoxaparin appeared to reduce the risk of CADVT by half. In post hoc analyses, reduction was limited to older children 1-17 years old. The goal of the CRETE Studies is to investigate this newly identified age-dependent heterogeneity in the efficacy of enoxaparin in reducing the risk of CADVT in critically ill children. To achieve this goal, the investigators aim (1) to confirm the efficacy and safety of early administration of prophylactic dose of enoxaparin in reducing the risk of CADVT in critically ill older children; (2) to determine the efficacy and safety of early administration of therapeutic dose of enoxaparin in reducing the risk of CADVT in critically ill infants; and, (3) to probe the mechanisms that underly the age-dependent heterogeneity in the efficacy of enoxaparin in reducing the risk of CADVT in critically ill children. The investigators will conduct 2 multicenter Bayesian explanatory randomized clinical trials in parallel to address Specific Aims 1 and 2. Depending on age, subjects will be randomized to different doses of enoxaparin vs usual care. Subjects will be systematically assessed for the development of CADVT using ultrasonography and clinically for bleeding. Using plasma obtained from subjects in the 2 trials, the investigators will conduct an exploratory mechanistic nested case-control study to address Specific Aim 3. Biomarkers of selected mechanisms underlying CVC-associated thrombus formation, particularly thrombin generation, will be compared between subjects with and without CADVT. The investigators will use Bayesian methods to improve the efficiency in the conduct and analyses of these studies. The CRETE Studies will provide high-quality age-appropriate evidence that will inform preventive strategies against CADVT and decrease harm in hospitalized children.

ELIGIBILITY:
Inclusion criteria

1. >36 weeks corrected gestational to <17 years old
2. <24 hours after insertion of an untunneled CVC
3. CVC inserted in the internal jugular or femoral vein

Exclusion criteria

1. Radiologic diagnosis of CADVT in the site of insertion in prior 6 weeks
2. Currently receiving an antithrombotic agent, e.g., LMWH, UFH, warfarin and aspirin, but not UFH at dose to maintain patency of a vascular catheter
3. Presence of clinically relevant bleeding, i.e., hemoglobin decreased ≥2 g/dl in 24 hours, required medical or surgical intervention to restore hemostasis, or in the retroperitoneum, pulmonary, intracranial or central nervous system, in the prior 60 days
4. Surgery in the prior 7 days
5. Major trauma in the prior 7 days
6. Presence of coagulopathy, i.e., INR >2.0, aPTT >50 seconds or platelet count <50 x 10^3/mcL
7. Presence of renal failure, i.e., creatinine clearance <30 mL/min/1.73 m2
8. Known hypersensitivity to heparin or pork products
9. Laboratory confirmed HIT
10. Current pregnancy or lactation
11. Presence of an epidural catheter
12. Limitation of care
13. Previous enrollment in the CRETE Studies

Max Age: 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 258 (Estimated)
Dates: Start 2022-05-11 (Actual); Primary Completion 2026-04-30 (Estimated); Study Completion 2026-07-31 (Estimated)

PRIMARY OUTCOMES:
Number of children with CADVT | Up to removal of CVC (maximum of 28 days)
  Thrombus in the central vein where the CVC was inserted that is diagnosed with systematic ultrasonographic surveillance.

SECONDARY OUTCOMES:
Number of children with any VTE | Up to removal of CVC (maximum of 28 days)
  Thrombus in the deep vein of any extremity or PE that is confirmed radiologically
Number of children with clinically apparent CADVT | Up to removal of CVC (maximum of 28 days)
  Any CADVT, except one that is only diagnosed with the systematic ultrasonographic surveillance.
Number of children with clinically apparent VTE | Up to removal of CVC (maximum of 28 days)
  Any VTE, except one that is only diagnosed with the systematic ultrasonographic surveillance.
Number of children with clinically relevant bleeding | Maximum of 36 hours after the last dose of enoxaparin
  Bleeding that is fatal, with drop in hemoglobin by ≥2 g/dl in 24 hours, requires medical or surgical intervention to restore hemostasis, or in the retroperitoneum, pulmonary or central nervous system.
Number of children with any bleeding | Maximum of 36 hours after the last dose of enoxaparin
  Any overt or macroscopic evidence of bleeding.
Number of children with heparin-induced thrombocytopenia | Maximum of 36 hours after the last dose of enoxaparin
  Unexplained drop in platelet count to <50 x 10^3/mcL or by 50 percent of baseline platelet count in the ICU within 21 days following exposure to heparin, and with a positive anti-platelet factor 4 antibody.

CONTACTS AND LOCATIONS:
Overall Officials: E. Vincent Faustino, MD, MHS, Principal Investigator — Associate Professor of Pediatrics, Yale School of Medicine
Locations (22):
- United States (22):
  - Children's of Alabama, Birmingham, Alabama
  - Arkansas Children's Hospital, Little Rock, Arkansas
  - Children's Hospital Colorado, Aurora, Colorado
  - Yale-New Haven Children's Hospital, New Haven, Connecticut
  - University of Florida -UF Health, Gainesville, Florida
  - Johns Hopkins All Children's, St. Petersburg, Florida
  - Children's Hospital of Illinois at OSF Saint Francis Medical Center, Peoria, Illinois
  - Stead Family Children's Hospital, Iowa City, Iowa
  - Children's Hospital St. Louis, St Louis, Missouri
  - Hassenfeld Children's Hospital, New York, New York
  - New York Presbyterian Hospital, New York, New York
  - Golisano Children's Hospital, Rochester, New York
  - Maria Fareri Children's Hospital, Valhalla, New York
  - UH Rainbow Babies & Children's Hospital, Cleveland, Ohio
  - Nationwide Children's Hospital, Columbus, Ohio
  - University of Oklahoma, Oklahoma City, Oklahoma
  - Penn State Hershey Children's Hospital, Hershey, Pennsylvania
  - Children's Hospital of Philadelphia, Philadelphia, Pennsylvania
  - Dell Children's Medical Canter, Austin, Texas
  - UTSW Medical Center; Children's Medical Center of Dallas, Dallas, Texas
  - Children's Hospital of Richmond, Richmond, Virginia
  - Children's Hospital Wisconsin, Milwaukee, Wisconsin

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Faustino EVS, Kandil SB, Leroue MK, Sochet AA, Kong M, Cholette JM, Nellis ME, Pinto MG, Chegondi M, Ramirez M, Schreiber H, Kerris EWJ, Glau CL, Kolmar A, Muisyo TM, Sharathkumar A, Polikoff L, Silva CT, Ehrlich L, Navarro OM, Spinella PC, Raffini L, Taylor SN, McPartland T, Shabanova V; Catheter-Related Early Thromboprophylaxis with Enoxaparin (CRETE) Studies Investigators and the Pediatric Critical Care Blood Research Network (BloodNet) of the Pediatric Acute Lung Injury and Sepsis Investigators Network (PALISI). Protocol for the Catheter-Related Early Thromboprophylaxis With Enoxaparin (CRETE) Studies. Pediatr Crit Care Med. 2025 Jan 1;26(1):e95-e105. doi: 10.1097/PCC.0000000000003648. Epub 2024 Nov 20. PMID 39560771